CLINICAL TRIAL: NCT00837382
Title: Imagery Rescripting for Posttraumatic Nightmares in Rural Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) Veterans With Posttraumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator is no longer a part of the VA.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Long, Mary - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24157
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Stress Disorders, Post-Traumatic; Sleep Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MEDVAMC Nightmare Treatment
  Interventions: Behavioral: MEDVAMC Nightmare Treatment
- 2 (Experimental): Videoconferencing nightmare Treatment
  Interventions: Behavioral: Telepsychiatry Nightmare Treatment

INTERVENTIONS:
Behavioral: MEDVAMC Nightmare Treatment — Veteran Nightmare Treatment Using Imagery Rescripting
  Arms: 1
Behavioral: Telepsychiatry Nightmare Treatment — Veteran Nightmare Treatment Using Imagery Rescripting Through Videoconferencing
  Arms: 2

SUMMARY:
Many service members returning from Iraq and Afghanistan have difficulties adjusting back to civilian life. Research shows that symptoms of posttraumatic stress disorder (PTSD) are particularly high in returning Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) veterans, and that combat-related nightmares and sleep disturbances are common in veterans with PTSD. This is of concern because people with these problems will often use unhealthy ways of coping. Although combat-related nightmares and difficulty sleeping are highly distressing, there are helpful treatments that do not involve taking medication. One of these treatments teaches specific skills to help people improve their sleep habits and to change their nightmares so that they are less upsetting. This treatment can be very helpful and research shows that people experience decreases in the frequency and severity of their nightmares, decreased symptoms of depression and PTSD, and improved sleep quality and quantity after completing treatment. However, because this treatment has only been studied with civilians, it is not clear how well this treatment works for returning veterans. This study tests how well this treatment works in treating combat nightmares in veterans who also have PTSD from experiencing a traumatic event.

ELIGIBILITY:
Inclusion Criteria:

Patients for the open trial will be

1. OEF/OIF veterans (aged 18-64);
2. English-speaking;
3. currently enrolled in the Trauma Recovery Program (TRP) at the Michael E. DeBakey Veteran Affairs Medical Center (MEDVAMC);
4. reporting at least one combat or war zone associated PTNM in the past week;
5. have an existing PTSD International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM); and
6. consenting to be in an open trial for treatment of PTNM. In addition, patients must agree to allow their assessment and therapy sessions to be video/audiotaped for the purposes of supervision.

Pilot Study: Patients for the pilot study will be

1. OEF/OIF veterans (aged 18-64);
2. English-speaking;
3. currently enrolled in the Conroe CBOC for their primary or mental health care;
4. reporting at least one combat or war zone associated PTNM in the past week;
5. have an existing PTSD ICD-9-CM diagnosis; and
6. consenting to be in the pilot study for treatment of PTNM. In addition, patients must agree to allow their assessment and therapy sessions to be video/audiotaped for the purposes of supervision.

Exclusion Criteria:

Patients will be excluded for the following reasons:

1. current active suicidal/homicidal ideation and intent;
2. current substance dependence;
3. a diagnosis of bipolar or psychosis;
4. active participation in another psychosocial treatment for PTSD;
5. prescribed the medication Prazosin (a psychotropic medication for the treatment of nightmares).

Patients interested in receiving the intervention will not be excluded if they are taking psychotropic medication (except for Prazosin) and may continue to take their medication as prescribed throughout the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS), Posttraumatic Stress Symptom Scale-Self-Report (PSS-SR) & Beck Depression Inventory-II (BDI-II) | Baseline & post-treatment

SECONDARY OUTCOMES:
Posttraumatic Cognitions Inventory (PTCI). | Baseline & post-treatment
The Pittsburgh Sleep Quality Index-Addendum for PTSD (PSQI) | Baseline & post-treatment
Trauma Related Nightmare Survey (TRNS). | Baseline & post-treatment
Mini-International Neuropsychiatric Interview (MINI) | Baseline
Treatment Evaluation Inventory (TEI) | Post-treatment
Client Satisfaction Questionnaire (CSQ) | Post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Long, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States